CLINICAL TRIAL: NCT02778347
Title: Development and Validation of a Comprehensive Standardised Clinical Assessment Tool for Patient Needs
Acronym: ACTI-PALLI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maison Médicale Jeanne Garnier (Other)
Collaborators: Ministère de la Santé (Unknown); Unité de Recherche Clinique Paris-Ouest (Unknown)
Responsible Party: Sponsor
Other Study IDs: 12-002-0105
Record Dates: First submitted 2015-01-08; First posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Palliative Care
Keywords: Palliative care; Need assessment; Tools; Validity; Quality of care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to develop and validate a comprehensive and standardised tool for assessment of patient needs in palliative care.

DETAILED DESCRIPTION:
Rationale for the study

In France, around 150000 people require palliative care every year. Since 2002, palliative care has been organized at several levels: palliative care units, palliative care mobile support teams, health network for palliative care and home-based hospital care. These structures have made possible for some patients in need of palliative care to be treated in appropriate service, in facility-based or community-based programs. With these important advances around palliative care, it appears important to assess the quality of care provided to patients. However, no generalizable study has been conducted in France, and no formal tool is available to help at this end.

In order to enhance the effectiveness of these services, it is important to conduct studies with the aim of developing the adapted and standardized tools that will enable assessment of quality for palliative care, as well as its determinants, for example the organization of structures, management of teams, etc. To this end, it is relevant to adopt a more holistic perspective and take into account the views of different concerned people, including the patients, their families and healthcare professionals, all while considering the organizational and management aspects.

The evidence from other countries has demonstrated the necessity of a rigorous, exhaustive and systematic evaluation as a requirement for any palliative program of quality. Many tools have since been developed to assess the multidimensional needs of patients, but none of these tools have been adapted to be used in the French palliative care settings.

Among of different tools used in palliative care, InterRAI Palliative Care (RAI-PC) has been chosen as the most reliable and complete tool. The RAI-PC allows a comprehensive evaluation of patients, as well as capabilities, preferences and needs. The medical, psychological, functional and social indicators are defined. This tool has been applied in the palliative care field in Canada and USA, but not yet in France. It has proven itself as an appropriate tool for needs assessment and evaluation of quality of care.

Goals of the project

This project aims to develop and validate a comprehensive and standardized instrument that will serve:

1. As a support to individual care, emphasizing the individual characteristics and needs of patients, informing planning care, outcome measurement, quality indicators, and case-mix classification.
2. As a standardized assessment tool adaptable to various palliative care structures

Study design

This study is a multicenter, prospective, observational study with representative stratified sample from different categories of palliative care services: palliative care units, palliative care mobile support teams, health network for palliative care and home-based hospital care. Twenty-three palliative structures, spread across the country are participating in this project.

The survey will involve the healthcare professionals of each center, trained on collecting information and using InterRAI instrument. Data collection involves patient clinical assessment, reviewing medical and nurse record and interview with family and professionals of healthcare.

Criteria for judgement

The quality of the tool will be judged in terms of satisfactory of psychometric properties, operational characteristics and clinical acceptability, adaptability of the tool to the needs of patients and its relevance in different palliative care structures.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women, age ≥ 18 years
* Patients receiving palliative care at home or in hospital at the time of screening

Exclusion Criteria:

* Non consenting
* Patient waiting a transfer within 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving palliative care
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Criterion-related validity: correlation between the score obtained using InterRAI-PC and scores obtained using MD Anderson Symptom Inventory (MDASI) | Baseline
  InterRAI-PC Scales versus MDASI scales (Pain Scale, dyspnea scale and Depression Rating Scale)

SECONDARY OUTCOMES:
Sensitivity to change: change in InterRAI-PC score over 7 days from Baseline | One Week
  InterRAI-PC scale
Inter-Observer Reliability of InterRAI-PC scale: correlation between score obtained by different observers (kappa coefficient) | Baseline
  InterRAI-PC scale

CONTACTS AND LOCATIONS:
Locations (1):
- Maison Médicale Jeanne Garnier, Paris, Paris, France